CLINICAL TRIAL: NCT02775032
Title: Evaluation of a Complex Intervention to Initiate Advance Care Planning in General Practice for the Improvement of End-of-life Care
Brief Title: Initiating ACP in General Practice. A Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Aline De Vleminck, Dr., Vrije Universiteit Brussel
Purpose: Health Services Research
Other Study IDs: VZP_HA_2016
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Life-threatening Illness; Palliative
Keywords: advance care planning; general practice; family practice; palliative care; end-of-life care

INTERVENTIONS:
Behavioral: Advance care planning conversations between patients and their GP

SUMMARY:
End-of-life care often fails in providing optimal patient-centred care and quality of life. Patients frequently suffer from inadequate control of pain, from a lack of communication about their illness and options for treatment, and from poor psychosocial and spiritual support. Advance care planning (ACP) can tackle these problems by providing patients with an opportunity to formulate their wishes and plan their future care, should they become incapable of participating in medical treatment decisions. Previous studies show that ACP improves concordance between patient's preferences and end-of-life care received and quality of care at the end-of-life. However, ACP is yet to be embedded in routine clinical practice and public consciousness. General practitioners (GPs) are in an ideal position to discuss ACP with their patients. By introducing ACP during a routine office visit, GPs can facilitate a structured discussion of the patient's wishes for end-of-life care. However, no ACP models have been systematically developed and tested in general practice. We developed a complex intervention to improve the initiation of ACP in general practice following the steps of an international guidance for development and evaluation of complex interventions. Before performing a full-scale intervention trial to study the effectiveness of this intervention on quality of care and quality of life, this model needs to be validated and tested in a pilot trial.

DETAILED DESCRIPTION:
Aim

1) to conduct the Phase II trial with GPs who will facilitate a structured ACP session with patients with a serious or life-threatening illness versus usual care and 2) to evaluate and validate the ACP intervention in terms of feasibility, acceptance to GPs and patients with a serious or life-threatening illness, and preliminary proof of effectiveness

Method

The implementation and preliminary evaluation of this intervention will be done by following the steps of the Medical Research Council (MRC) framework on complex intervention designs. This framework proposes a stepwise approach going from phase 0 to phase IV.

Phase 0-I were previously conducted by the research team and comprised the development of the intervention. This project proposal comprises phase II (exploratory trial) in which the feasibility and acceptability of the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with a serious or life-threatening illness
* older than 18 years
* Dutch speaking
* eligible according to the Surprise question
* able to give informed consent
* able to complete questionnaires and participate in qualitative interview

Exclusion Criteria:

* younger than 18 years
* incompetent to participate due to mental incapacity
* unable to give informed consent
* unable to complete questionnaires or participate in qualitative interviews

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire | up to 1 month

REFERENCES:
- [Derived] Dierickx S, Pardon K, Pype P, Stevens J, Vander Stichele R, Deliens L, De Vleminck A. 'Advance care planning, general practitioners and patients: a phase II cluster-randomised controlled trial in chronic life-limiting illness'. BMJ Support Palliat Care. 2020 Dec 2:bmjspcare-2020-002712. doi: 10.1136/bmjspcare-2020-002712. Online ahead of print. PMID 33268475